CLINICAL TRIAL: NCT00388622
Title: Improving Drug Use for Elderly Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Indiana University School of Medicine (Other); Purdue University (Other); Wishard Health Services (Other)
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01AG019105 (NIH)
Record Dates: First submitted 2006-10-08; First posted 2006-10-17 (Estimated); Last update posted 2006-10-17 (Estimated); Status verified 2006-10

CONDITIONS: Heart Failure
Keywords: Heart failure; Adherence; Compliance; Pharmacy; Pharmacist; Health-related quality of life; Clinical exacerbation; Costs
MeSH Terms: conditions — Heart Failure; Patient Compliance

INTERVENTIONS:
Behavioral: Pharmacist intervention

SUMMARY:
The aims of this randomized, clinical trial are to develop and test a multileveled pharmacy-based program to improve the care of patients with heart failure. Risk factors for deterioration of heart failure will be determined including poor adherence to medication.

DETAILED DESCRIPTION:
Medications improve the function and health-related quality of life of patients with heart failure and reduce morbidity, mortality, and the costs of patient care. Due to their complicated medication regimens, however, older adults with heart failure require assistance with their medications to facilitate adherence and improve their health outcomes. Recent studies suggest that the outcomes of patients with heart failure improve when pharmacists provide patients with education and monitoring. This study aims to develop and test, as a randomized controlled trial, a multileveled pharmacy-based program that incorporates patient education materials and medication packaging that target patients with low health literacy.

Elderly patients from Wishard Health Services with a diagnosis of heart failure (n=314) were randomly assigned to the pharmacist intervention or usual care group. Patients in the intervention group received verbal and written education, icon-based labeling of their medication containers, and therapeutic monitoring. A main objective of the pharmacist was to reinforce primary care providers' instructions to the patient. The pharmacist educated patients about their medications, identified barriers to appropriate drug use, coached patients on overcoming drug use barriers, and coordinated drug use for these patients with primary care providers. Patients in the usual care (control) group did not receive the intervention and also served as a prospective cohort to identify the determinants of acute exacerbation.

To measure medication compliance objectively, electronic monitor lids were used on all heart failure medications for patients in intervention and control groups. These lids contain a computer chip that electronically imprints a time/date stamp when opened and closed. Each open-close event indicates that the patient has taken a dose of their medication. By downloading this information from the medication container lid to a computer, we can objectively assess the pattern of medication compliance. Study participation for the patients in the intervention group concluded after nine months of active intervention and three months of post-intervention follow-up.

The usual care group permitted our identification of the causes for clinical deterioration in patients with heart failure. The unique electronic medical record at our institution, the Regenstrief Medical Record System, permits capture of a wealth of clinical data, which can be merged with primary data from the trial (for example, medication adherence by MEMS caps, brain natriuretic peptide, and quality of life assessments). Patients' data captured from the Regenstrief Medical Record System during the year of follow-up were used to perform multivariate analyses to determine causes of clinical deterioration. So doing provided insights into the pathophysiology of decompensation in patients with heart failure to enhance our understanding of risk factors of this increasingly prevalent disease and thereby lead us to better therapeutic strategies.

Covariates used in our analyses of risk factors included age, sex, race, weight, ejection fraction, brain natriuretic peptide and other renal autacoids, and New York Heart Association classification. Endpoints include health-related quality of life, heart failure exacerbation, patient satisfaction, and healthcare costs. We evaluated the effectiveness of the pharmacy-based program in improving adherence to heart failure medications, improving health-related quality of life, decreasing heart failure exacerbations, increasing patient satisfaction, and decreasing health care costs. Once identified, factors predicting decompensation of heart failure may become the targets of future interventions aimed at preventable causes.

ELIGIBILITY:
Inclusion Criteria:

* age 50 and older
* prescription for at least one cardiovascular medication for heart failure
* plan to receive care and prescriptions at the study health care facility
* ability to hear within the normal range of conversation
* English speaking
* willingness to obtain echocardiography

Exclusion Criteria:

* dementia

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314
Dates: Start 2001-02; Study Completion 2004-11

PRIMARY OUTCOMES:
Medication adherence
Exacerbation of heart failure
Health-related quality of life

SECONDARY OUTCOMES:
Patient satisfaction
Health care utilization
Direct costs

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Murray, PharmD, MPH, Principal Investigator — UNC-Chapel Hill
Locations (1):
- UNC Chapel Hill, School of Pharmacy, CB 7360, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Noureldin M, Plake KS, Morrow DG, Tu W, Wu J, Murray MD. Effect of health literacy on drug adherence in patients with heart failure. Pharmacotherapy. 2012 Sep;32(9):819-26. doi: 10.1002/j.1875-9114.2012.01109.x. Epub 2012 Jun 28. PMID 22744746
- [Derived] Kim KM, Murray MD, Tu W, Robarge J, Ding Y, Brater DC, Flockhart DA. Pharmacogenetics and healthcare outcomes in patients with chronic heart failure. Eur J Clin Pharmacol. 2012 Nov;68(11):1483-91. doi: 10.1007/s00228-012-1280-z. Epub 2012 Apr 29. PMID 22543981
- [Derived] Murray MD, Ritchey ME, Wu J, Tu W. Effect of a pharmacist on adverse drug events and medication errors in outpatients with cardiovascular disease. Arch Intern Med. 2009 Apr 27;169(8):757-63. doi: 10.1001/archinternmed.2009.59. PMID 19398687
- [Derived] Murray MD, Tu W, Wu J, Morrow D, Smith F, Brater DC. Factors associated with exacerbation of heart failure include treatment adherence and health literacy skills. Clin Pharmacol Ther. 2009 Jun;85(6):651-8. doi: 10.1038/clpt.2009.7. Epub 2009 Mar 4. PMID 19262464
- [Derived] Murray MD, Young J, Hoke S, Tu W, Weiner M, Morrow D, Stroupe KT, Wu J, Clark D, Smith F, Gradus-Pizlo I, Weinberger M, Brater DC. Pharmacist intervention to improve medication adherence in heart failure: a randomized trial. Ann Intern Med. 2007 May 15;146(10):714-25. doi: 10.7326/0003-4819-146-10-200705150-00005. PMID 17502632